CLINICAL TRIAL: NCT06610760
Title: Efficacy and Safety of Ursodeoxycholic Acid in Reversing Gastric Intestinal Metaplasia: A Multicenter, Randomized, Placebo-Controlled Trial
Brief Title: Efficacy and Safety of Ursodeoxycholic Acid in Reversing Gastric Intestinal Metaplasia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yongquan Shi (Other)
Responsible Party: Sponsor-Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20242225-F-1
Record Dates: First submitted 2024-09-19; First posted 2024-09-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-07

CONDITIONS: Gastric Intestinal Metaplasia
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The ursodeoxycholic acid group (Experimental): Patients in the ursodeoxycholic acid group will receive oral ursodeoxycholic acid at a dosage of 250 mg three times daily for 6 months.
  Interventions: Drug: Ursodeoxycholic Acid
- The placebo group (Placebo Comparator): Patients in the placebo group will receive oral placebo at a dosage of 250 mg three times daily for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Subjects will be instructed to take one capsule (250mg) of ursodeoxycholic acid three times daily, and visit the hospital every 4 weeks for evaluation of the subjective symptoms and to receive a new supply of medication.
  Arms: The ursodeoxycholic acid group
Drug: Placebo — Subjects will be instructed to take one capsule (250mg) of placebo three times daily, and visit the hospital every 4 weeks for evaluation of the subjective symptoms and to receive a new supply of medication.
  Arms: The placebo group

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of ursodeoxycholic acid in treating gastric intestinal metaplasia in Helicobacter pylori-negative adults. It will also learn about the safety of ursodeoxycholic acid. The main questions it aims to answer are:

Does ursodeoxycholic acid promote the regression of IM in individuals without Helicobacter pylori infection? What medical problems do participants experience when taking ursodeoxycholic acid? Researchers will compare ursodeoxycholic acid to a placebo (a look-alike substance that contains no drug) to see if ursodeoxycholic acid is effective in treating gastric intestinal metaplasia.

Participants will:

Take ursodeoxycholic acid or a placebo every day for 6 months. Visit the clinic once every 4 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 to 75 years old.
* patients with OLGIM stage Ⅱ-Ⅳ diagnosed by upper gastrointestinal endoscopy and histopathological examination within the last 3 months.
* patients without Helicobacter pylori infection, including patients who had successful Helicobacter pylori eradication before enrollment.

Exclusion Criteria:

* a history of regular use (defined as at least once per week) of non-steroidal anti-inflammatory drugs (NSAIDs) and/or statins.
* a history of stomach surgery (including endoscopic submucosal dissection and endoscopic mucosal resection) or previously diagnosed malignant tumor.
* a history of heart failure, renal failure, liver cirrhosis or chronic hepatic failure; patients with contraindications or allergies to the drugs in this study.
* breastfeeding or pregnancy.
* a history of substance abuse or alcohol abuse within the past one year.
* patients with severe mental illness.
* refusal to undergo drug treatment.
* refusal to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The regression rate of gastric intestinal metaplasia based on OLGIM stage in different groups. | From enrollment to the end of treatment at 6 months
  Regression was defined as a OLGIM stage decreased at least one grade.
The progression rate of gastric intestinal metaplasia based on OLGIM stage in different groups. | From enrollment to the end of treatment at 6 months
  Progression was defined as a OLGIM stage increased at least one grade.

SECONDARY OUTCOMES:
The regression rate of gastric atrophy based on OLGA stage in different groups. | From enrollment to the end of treatment at 6 months
  Regression was defined as a OLGA stage decreased at least one grade.
The progression rate of gastric atrophy based on OLGA stage in different groups. | From enrollment to the end of treatment at 6 months
  Progression was defined as a OLGA stage increased at least one grade.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, PhD, Study Chair — Air Force Military Medical University, China; Xinzhao Wang, Principal Investigator — 989 Hospital of PLA Joint Logistics Support Force; Kun Zhuang, Principal Investigator — Xi'an Central Hospital; Zhufang Ma, Principal Investigator — Hanzhong 3201 Hospital; Yuan Gao, Principal Investigator — Ankang Central Hospital; Long Zou, Principal Investigator — Shangluo Central Hospital
Locations (6):
- China (6):
  - 989 Hospital of PLA Joint Logistics Support Force, Pingdingshan, Henan
  - Ankang Central Hospital, Ankang, Shaanxi
  - Hanzhong 3201 Hospital, Hanzhong, Shaanxi
  - Shangluo Central Hospital, Shangluo, Shaanxi
  - Xijing hospital, Xi'an, Shaanxi
  - Xi'an Central Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No